CLINICAL TRIAL: NCT03703206
Title: The Analgesic Efficacy of Adding the IPACK Block to a Multimodal Analgesia Protocol for Primary Total Knee Arthroplasty
Brief Title: The Analgesic Efficacy of Protocol for Primary Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 828618
Record Dates: First submitted 2018-07-27; First posted 2018-10-11 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, blinded study with a parallel design and an allocation ratio of 1 to 1 for the treatment groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ACB + iPACK (Experimental): Patients scheduled for TKA will be randomized to receive an adductor canal block with an additional ultrasound guided injection of local anesthetic between the popliteal artery and the capsule of the knee (iPACK).
  Interventions: Drug: ultrasound guided injection of local anesthetic between the popliteal artery and the capsule of the knee (iPACK)
- ACB w/o iPACK (No Intervention): Patients enrolled in this arm will receive the standard of care adductor canal block (ACB) prior to their total knee arthoplasty.

INTERVENTIONS:
Drug: ultrasound guided injection of local anesthetic between the popliteal artery and the capsule of the knee (iPACK) — nerve block for posterior knee pain after a TKA.
  Other Names: iPACK
  Arms: ACB + iPACK

SUMMARY:
This is a perspective, randomized, blinded study with a parallel design and an allocation ratio of 1 to 1 for the treatment groups to assess the analgesic efficacy of adding the iPACK (injection between the popliteal artery and the capsule of the knee) in addition to the adductor canal block (ACB) for Total Knee Arthoplasty patients (TKA).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty
* American Society Anesthesiologists (ASA) physical status I- III.
* Mentally competent and able to give consent for enrollment in the study.

Exclusion Criteria:

* Patient refusal,
* allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone, and any of the drugs included in the multimodal perioperative pain protocol (MP3).
* Revision surgery will be excluded.
* Impaired kidney functions
* patient with coagulopathy will be also excluded.
* Chronic pain syndromes and patients with chronic opioid use in excess of a daily morphine equivalent dose (MED) of 40mg or greater for the past 3 months prior to the surgery.
* BMI of 45 or more

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taras Grosh, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four hundred and sixty-four patients were screened for eligibility, with 120 patients ultimately enrolling in the study. Of the 120 patients enrolled, 119 patients completed all necessary follow-up for inclusion into the study
Pre-assignment Details: 120 patients enrolled, 119 patients completed all necessary follow-up for inclusion in the study: 60 patients in the IPACK group and 59 patients in the sham group. There were no block failures. These 119 patients were randomized to receive either an IPACK or a sham block in addition to multimodal analgesia and an ACB. We were set to assess pain in the back of the knee 6 hours after surgery, quality of recovery after surgery, pain scores, opioid requirements, and functional measures
Period: Overall Study
Arm/Group | ACB + iPACK | ACB w/o iPACK
Started | 60 | 59
Completed | 60 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACB + iPACK | ACB w/o iPACK | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: Age (years)] | 67.7 (7.8) | 65.6 (8.2) | 66.7 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 26 | 24 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 38 | 83
  African American | 14 | 20 | 34
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Presenting With Pain in the Back of the Knee 6 Hours After Surgery
Description: Each patient will be provided by a colored chart that will have different parts of the knee marked clearly and they will indicate whether the pain they have in which region of the knee. the different regions are ( anterior, posterior, lateral, medial, and the middle of the thigh). it will be marked as a yes or no question. it will be measured as a ratio of patients in each patient who has the pain in the numerator and all patients in the study will be in the denominator
Time Frame: Six hours after surgery
Measure: Number; unit: percentage of patients reporting pain
Arm/Group | ACB + iPACK | ACB w/o iPACK
Number analyzed (Participants) | 60 | 59
percentage of patients reporting pain | 21.7 | 45.8

2. Secondary Outcome: Pain Score Measurement Reported by Patients
Description: Average of pain scores over the first 24 hours following the regional anesthetic based on Numeric Rating Scale ( NRS). The scale is from 0 - 10, where 0 is no pain and 10 is the worst pain possible.
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: pain scores
Arm/Group | ACB + iPACK | ACB w/o iPACK
Number analyzed (Participants) | 60 | 59
pain scores | 5 (0.01) | 6 (0.01)

3. Secondary Outcome: Quality of Recovery (QoR) Score
Description: Score of QoR-15 survey to determine recovery status. The questionnaire is a 15 item questionnaire and each question has a score possible from 0-10. It has two parts. Part 1 includes questions from 1-10. the scale on this question ranges from 0=none of the time ( poor) to 10=all the time ( excellent). The 2nd part include questions from 11-15 where the scale goes from 10 to 0, where 10=none of the time ( excellent) and 0=all the time (poor). The total score is obtained by adding the scores of all the 15 questions. The total score is 0 (poor_ to 150 (excellent).
Time Frame: one week, measurements are obtained at 24 hours, 48 hours, and one week
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | ACB + iPACK | ACB w/o iPACK
Number analyzed (Participants) | 60 | 59
score on a scale
  Postoperative Day 1 | 113 (0.66) | 114 (0.66)
  Postoperative Day 2 | 118 (0.37) | 123 (0.37)
  Postoperative Day 7 | 131 (0.11) | 126 (0.11)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | ACB + iPACK | ACB w/o iPACK
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03703206/Prot_SAP_000.pdf